CLINICAL TRIAL: NCT04886037
Title: The Sestrin Levels in Patients With Endometriosis
Brief Title: Evaluation of Sestrin Levels in Patients With Endometriosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Yalcin bahat, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: endo-sestrin
Record Dates: First submitted 2021-05-09; First posted 2021-05-13 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis
Keywords: sestrin
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with endometriosis: It consists of women between the ages of 18-45 who have been diagnosed with endometriosis by surgery or ultrasonography.
  Interventions: Other: sestrin
- control: It consists of healty women between the ages of 18-45
  Interventions: Other: sestrin

INTERVENTIONS:
Other: sestrin — Serum sestrin levels involved in inflammation and energy metabolism are compared between endometriosis and healthy control group.

SUMMARY:
Serum sestrin levels of endometriosis patients are compared with a group of healthy volunteers of the same age.

DETAILED DESCRIPTION:
Serum sestrin levels are compared with 45 endometriosis patients and 45 healthy volunteers of the same age. The energy metabolism of the endometriosis group and its possible relationship with the endometriosis stage will be compared since sestrin gives information about the energy metabolism of the people.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with endometriosis (Surgery or ultrasound)
* Women without endometriosis

Exclusion Criteria:

* Women without endometriosis
* women who are only suspected endometriosis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: The serum sestrin level of women between the ages of 18-45 who have been diagnosed with endometriosis by surgery or ultrasound will be compared with the level of women of the same age.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-10 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Serum sestrin levels in women with endometriosis | 6 months
  Serum sestrin levels involved in inflammation and energy metabolism are compared between endometriosis and healthy control group.

SECONDARY OUTCOMES:
Comparison of the relationship between serum sestrin level and endometriosis stage | 6 months
  By comparing the relation of serum sestrin level with the stage of endometriosis, its relation with serum level in patients with advanced and early stage endometriosis will be examined. The possible effect of sestrin on disease pathogenesis will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Pinar Yalcin Bahat, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided